CLINICAL TRIAL: NCT05810337
Title: The Effects of Splenda (Sucralose) on Blood Glucose Concentration, Appetite Scores and Subsequent Energy Intake in Humans: a Randomised Controlled Trial
Brief Title: Splenda: Effects on Blood Glucose Concentration, Appetite Scores and Subsequent Energy Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Dr Christopher Corpe, Nutrition Sciences Lecturer, Principal investigator, King's College London
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: KCLMScNutr2023
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Appetitive Behavior; Glucose Metabolism Disorders
Keywords: Blood glucose; Appetite; Energy intake
MeSH Terms: conditions — Appetitive Behavior; Glucose Metabolism Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Splenda drink (Experimental): Drink containing 4.5g Splenda dissolved on 250ml water.
  Interventions: Dietary Supplement: Splenda drink; Dietary Supplement: High carbohydrate breakfast
- Maltodextrin drink (Placebo Comparator): Drink containing 4.5g maltodextrin dissolved on 250ml water.
  Interventions: Dietary Supplement: Maltodextrin drink; Dietary Supplement: High carbohydrate breakfast

INTERVENTIONS:
Dietary Supplement: Splenda drink — 4.5g Splenda containing 1% sucralose, 95% maltodextrin, dissolved in 250ml water and consumed with a high carbohydrate breakfast.
  Arms: Splenda drink
Dietary Supplement: Maltodextrin drink — 4.5g maltodextrin dissolved in 250ml water and consumed with a high carbohydrate breakfast.
  Arms: Maltodextrin drink
Dietary Supplement: High carbohydrate breakfast — Meal consisting of 30g cereal with 100ml skimmed milk, 1.5 slices white toast with 12g margarine, providing 386kcal, 61.4g carbohydrate, 10.4g protein and 10.1g fat.

SUMMARY:
This study investigates the effects of Splenda, an artificial sweetener powder containing sucralose, on post-prandial blood glucose levels, appetite scores and subsequent energy intake.

DETAILED DESCRIPTION:
Participants are randomly assigned to receive either the placebo drink (4.5g maltodextrin dissolved in 250ml water) or the Splenda drink (4.5g Splenda dissolved in 250ml water) taken alongside a high calorie breakfast.

Blood glucose measurements will be obtained through finger-pricking and appetite will be measured using self-reported visual analogue scores rating hunger, desire to eat, fullness and alertness for up to 3 hours after breakfast. Energy intake will be measured using a 24 hour food diary.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults (18-64 years)

Exclusion Criteria:

-

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Change in blood glucose | -5 to 180 minutes (measured from baseline up to 90min every 15min and from 90-180min every 30min)
  Capillary blood glucose from fingerprick and measured using glucose monitor
Change in appetite | -5 to 180 minutes (measured from baseline up to 90min every 15min and from 90-180min every 30min)
  Feelings of hunger, desire to eat, fullness and alertness measured using Visual Analogue Scale (VAS)

SECONDARY OUTCOMES:
24 hour energy intake | 0 - 24 hours
  Food intake over the 24 hours of the study day using a 24 hour food diary entered into dietary analysis software

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Corpe, Dr., Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No